CLINICAL TRIAL: NCT00005164
Title: Insulin Resistance and Blood Pressure Regulation in Blacks
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1036; R01HL031802 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Hypertension; Heart Diseases; Insulin Resistance
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Heart Diseases; Insulin Resistance

SUMMARY:
To determine the role of insulin resistance in peripheral vascular dynamics, sodium sensitivity, and blood pressure regulation in a young representative Black population and in a group of young Blacks at high risk for hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

Epidemiologic studies have demonstrated a greater prevalence of essential hypertension in Blacks with a disproportionately greater hypertension related mortality in Blacks. Similar vascular consequences occur with diabetes and obesity. These three diseases not only share a common outcome, but also overlap in occurrence with Blacks having greater prevalence rates in the three disorders. Insulin resistance has been documented in all three disorders and may contribute significantly to the vascular disease.

This project originated in response to a Request for Applications on Biobehavioral Factors Affecting Hypertension in Blacks issued in December 1982. The original project was supported by the RFA for three years. The first three years of the study focussed on the hypothesis that sodium loading would augment cardiovascular responses of psychogenic stress in Blacks at high risk for hypertension. The first phase of the study examined and compared 80 Blacks and whites, 18-22 years of age. The second phase involved an additional 40 Black borderline hypertensives who were exposed to the same set of studies designed to examine possible interactions between neurogenic and renal controlled volume mechanisms in essential hypertension.

The project was renewed as a regular research grant in 1986 and was designed to investigated biobehavioral factors in blood pressure control. In 1988, the study on insulin resistance was funded and continued through 1990.

DESIGN NARRATIVE:

Subjects in this project consisted of Blacks who were enrolled in the Collaborative Perinatal Project (CPP) at birth and who had been studied longitudinally in adolescence and young adulthood. Each subject brought to the study data on blood pressure, growth, and maturation from birth through late adolescence.

Peripheral vascular structure was studied using measures of forearm blood flow and forearm vascular resistance. Measurements of peripheral vascular structure were compared to data on sodium sensitivity and potassium sensitivity in the population. Insulin resistance was studied using the euglycemic hyperinsulinemic clamp technique. Variations in the activity of the sodium-potassium pump and sodium-hydrogen exchange in red cells were correlated with insulin resistance to determine if hyperinsulinemia alters cation transport rates.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1983-09; Study Completion 1991-08 (Actual)

REFERENCES:
- [Background] Canessa M, Spalvins A, Adragna N, Falkner B. Red cell sodium countertransport and cotransport in normotensive and hypertensive blacks. Hypertension. 1984 May-Jun;6(3):344-51. doi: 10.1161/01.hyp.6.3.344. PMID 6735456
- [Background] Chinese M, Solomon H, Falkner B, Adragna N, Ellison RC: Familial Aggregation of Sodium Countertransport and Cotransport and Essential Hypertension in: Topics on Pathophysiology of Hypertension. Villareal H, Sambhi MP, Nijhoff Publish. Boston, p. 78-87, 1984
- [Background] Falkner B, Katz S, Chinese M, Kushner H: The Response to Chronic Oral Sodium Loading in Young Blacks. Hypertension, 8 (Suppl I): I-165-168, 1986
- [Background] Falkner B. Cardiovascular characteristics of the young with borderline hypertension. J Cardiovasc Pharmacol. 1986;8 Suppl 5:S44-7. doi: 10.1097/00005344-198608005-00009. PMID 2427884
- [Background] Canessa M, Bize I, Spalvins A, Falkner B, Katz S. Na-K-C1 cotransport and Na pump in red cells of young blacks and blood pressure response to salt loading. J Clin Hypertens. 1986 Jun;2(2):101-8. PMID 2428944
- [Background] Falkner B, Ragonesi S. Psychosocial stress and reactivity as risk factors of cardiovascular disease. J Am Acad Child Psychiatry. 1986 Nov;25(6):779-84. doi: 10.1016/s0002-7138(09)60195-3. No abstract available. PMID 3794120
- [Background] Falkner B, Light K: The Interactive Effects of Stress and Dietary Sodium on Cardiovascular Reactivity. In: J Hypertens, Stress, Reactivity, and Cardiovascular Disease: Status and Prospects. Eds. Matthews L, Weiss SM, Detre T, Dembroski T, Falkner B, Manuch S, Williams R (Eds), John Wiley and Sons, Inc. New York, p 329-341, 1986
- [Background] Falkner B: Mild Hypertension in Adolescence. In: Mild Hypertension: From Drug Trials to Practice. Strasser T, Gaten D, (Eds) Raven Press, New York, p 279-283, 1987
- [Background] Falkner B, Kushner H, Khalsa DK, Canessa M, Katz S. Sodium sensitivity, growth and family history of hypertension in young blacks. J Hypertens Suppl. 1986 Dec;4(5):S381-3. PMID 3471912
- [Background] Falkner B: Reactivity to Mental Stress in Hypertension and Prehypertension in: Handbook of Hypertension, Vol. 10. Behavioral Factors in Hypertension, Editor Julius S. and Bassett DR. Elsevier Science Publishers. B.V., 1987
- [Background] Falkner B. Sodium sensitivity: a determinant of essential hypertension. J Am Coll Nutr. 1988 Feb;7(1):35-41. doi: 10.1080/07315724.1988.10720218. PMID 3278039
- [Background] Falkner B: Measurement of Volume Regulation: Renal Function. in: Schneiderman N, Kaufman P and Weiss SM (Eds). Handbook of Research Methods in Cardiovascular Behavioral Medicine. New York: Plenum Publishing Corporation, 1989
- [Background] Falkner B. Vascular reactivity and hypertension in childhood. Semin Nephrol. 1989 Sep;9(3):247-52. No abstract available. PMID 2675243
- [Background] Santangelo K, Falkner B, Kushner H. Forearm hemodynamics at rest and stress in borderline hypertensive adolescents. Am J Hypertens. 1989 Jan;2(1):52-6. doi: 10.1093/ajh/2.1.52. PMID 2914085
- [Background] Falkner B, Kushner H. Race differences in stress-induced reactivity in young adults. Health Psychol. 1989;8(5):613-27. doi: 10.1037//0278-6133.8.5.613. PMID 2630296
- [Background] Falkner B, Kushner H. Effect of chronic sodium loading on cardiovascular response in young blacks and whites. Hypertension. 1990 Jan;15(1):36-43. doi: 10.1161/01.hyp.15.1.36. PMID 2295513
- [Background] Falkner B. Differences in blacks and whites with essential hypertension: biochemistry and endocrine. State of the art lecture. Hypertension. 1990 Jun;15(6 Pt 2):681-6. doi: 10.1161/01.hyp.15.6.681. PMID 2190920
- [Background] Falkner B, Hulman S, Tannenbaum J, Kushner H. Insulin resistance and blood pressure in young black men. Hypertension. 1990 Dec;16(6):706-11. doi: 10.1161/01.hyp.16.6.706. PMID 2246037
- [Background] Canessa M, Laski C, Falkner B. Red blood cell Na+ transport as a predictor of blood pressure response to Na+ load in young blacks and whites. Hypertension. 1990 Nov;16(5):508-14. doi: 10.1161/01.hyp.16.5.508. PMID 2228151
- [Background] Falkner B: Etiologic Factors in Essential Hypertension. Loggie J, Robson A (Eds), in: Pediatric and Adolescent Hypertension, 1992.
- [Background] Falkner B, Rabinowitz AI, Michel SH: Nutrition and Blood Pressure in Childhood: In: Nutritional Factors in Hypertension, Langford H, Levine B (Eds), Alan R Liss, Inc., New York, 1990.
- [Background] Falkner B, Kushner H. Interaction of sodium sensitivity and stress in young adults. Hypertension. 1991 Jan;17(1 Suppl):I162-5. doi: 10.1161/01.hyp.17.1_suppl.i162. PMID 1986997